CLINICAL TRIAL: NCT03581721
Title: Prevention of Maternal Hypothermia After Scheduled Caesarean Section Using Active IV Fluid Warming: a Randomized Controlled Trial
Brief Title: Prevention of Maternal Hypothermia After Scheduled Caesarean Section Using Active Intravenous Warming
Acronym: CESAR-RESOL2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K170402J; 2017-A03139-4 (Registry Identifier: ANSM)
Record Dates: First submitted 2018-04-05; First posted 2018-07-10 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Hypothermia
Keywords: Postoperative hypothermia; caesarean section; IV fluids warming

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (No Intervention): Control group according to usual practices: no active warming (no fluid warming). The fluid warmer device will be set up but not activated. The control group will receive IV fluid coload at room temperature through the fluid warmer set to "off". The device is hidden
- The warming group (Experimental): "IV fluid warming with the enFlow® or Fluido®Compact IV fluid warmer" : Women will receive IV fluid coload warmed to 40°C through the enFlow® or Fluido®Compact device. The box will be also hidden. The fluid warmer will be turned off at the end of surgery, just before transfer to the PACU.
  Interventions: Device: enFlow® IV fluid warmer and from July 2019 Fluido®Compact IV fluid warmer

INTERVENTIONS:
Device: enFlow® IV fluid warmer and from July 2019 Fluido®Compact IV fluid warmer — The fluid warmer will be set up by an external co-investigator in every patient included in the study. It will be turned on in patients belonging to the "warming" group, and turned off in the control group
  Arms: The warming group

SUMMARY:
Maternal hypothermia is very frequent after caesarean delivery under spinal anaesthesia and should be prevented, as it induces discomfort and increases the risk of postoperative complications. Several modalities of active warming have been explored, with contrasting results. Small IV Fluid warming systems offer effective and safe IV fluid warming without discomfort, and are very easy to use. The investigators hypothesize that such devices can efficiently prevent hypothermia after caesarean section even with high flow rates of infusion. The purpose of this study is to determine whether active fluid warming reduces the occurrence of maternal hypothermia after scheduled caesarean section, as compared with no active warming. The investigators plane to conduce a double-blinded randomized controlled trial. Seventy women undergoing scheduled caesarean section under spinal anaesthesia in 3 different maternity units will be included. The primary outcome is the occurrence of maternal hypothermia (<36.0°C) on admission to the post anaesthesia care unit. The secondary outcomes are perioperative maternal hypothermia, maternal thermal discomfort, maternal recovery and neonatal well-being

DETAILED DESCRIPTION:
Hypothermia is a well-known complication of general and neuraxial anaesthesia. After a caesarean section under spinal anaesthesia, 30 to 40% of the mothers have a core temperature <36°C. Perioperative hypothermia induces maternal thermal discomfort and shivering, but also increases the amount of blood loss and the risks of postoperative wound infections and cardiac complications. In addition, maternal hypothermia may also have an impact on neonatal outcomes. Prevention of maternal hypothermia in women scheduled for caesarean delivery is consequently necessary, and is an important part of enhanced recovery after surgery. Active warming is efficient in preventing postoperative hypothermia. Forced-air warming is the most commonly used modality of active warming. However forced-air warming should be applied for at least 60 minutes to be efficient. As surgical duration for a caesarean is lower than one hour, this technic does not appear really appropriate in this context. In addition, upper body forced-air warming is uncomfortable for women and can interfere with bonding. Consequently forced-air warming is not generally used during caesarean delivery. Warmed IV fluid is another option to prevent perioperative hypothermia, but with contrasting results, depending mainly on the device and on the amount of perioperative fluids infusion. Co-loading IV fluid is recommended to prevent maternal hypotension induced by spinal anaesthesia in the context of caesarean delivery. Small released fluid warmings routinely used in scheduled surgery, are able to warm IV fluid administered with high flows, such as in co-loading IV fluid. But the efficiency of these devices to prevent maternal hypothermia has never been explored in the context of caesarean section under spinal anaesthesia with co-loading.

The investigators hypothesized that warmed IV fluid administered in co-loading with enFlow® or Fluido®Compact decreases the incidence of postoperative maternal hypothermia after caesarean section under spinal anaesthesia.

The investigators will perform a double blinded randomized controlled trial comparing active IV warming with enFlow® or Fluido®Compact versus placebo.

Indeed at the beginning of the study, the performance of the enFlow device were tested. But in February 2019, a study published in Anaesthesia showed that uncoated aluminium plates in fluid warming systems, such as those used in the enFlow system, yielded potentially harmful concentrations of aluminium when using balanced electrolyte solutions (ref Perl Anaesthesia 2019). Consequently this device was quarantined unless there are no alternative fluid warmers available Of note no adverse event has been reported associated with the use of enFlow® device. Consequently, we choose to continue our study with the Fluido®Compact, which is a very similar small fluid warmer but with coated aluminium plate.

After obtaining written informed consent from the patients, 70 pregnant women ASA status 1 or 2 and scheduled for caesarean delivery will be enrolled and randomized into two groups: active IV fluid warming vs no active warming. Written informed consent will be obtained before randomisation using an Internet based randomisation system. Participants will be randomized just after their arrival in the operative room. The clinicians in charge of the patients, the researcher and the woman will be blinded. In the operative room, a venous cannula will be inserted into the forearm, and an infusion of Ringer's lactate solution fluids will be initiated. An enFlow® or Fluido®Compact device will be placed on the IV for all the patients, but turned on only in the group active warming. The device will be hidden in all the patients. Every patient will have a spinal anaesthesia in sitting position with hyperbaric bupivacaine 10mg, sufentanil 3µg and morphine 100µg. An IV co loading with Ringer-Lactate 1000 ml will be started at the beginning of the spinal administration. All the women will be monitored using heart rate, continuous SpO2, non-invasive arterial blood pressure every 1-minute until the baby is born, and then every 5 minutes. Maternal arterial hypotension will be corrected with ephedrine or phenylephrine as appropriate. All the women will receive carbetocin 100µg just after baby extraction. While in the operative room, all the data will be collected on a standardized data collection sheet. In case of maternal temperature <35°C during surgery, an active warming blanket will be used. The enFlow® or Fluido®Compact device will be taken off at the end of the surgery just before leaving the operative room.

In addition, postoperative data will be collected during the admission to the post-anaesthesia care unit (PACU). In case of maternal temperature <36°C in the PACU, a warming blanket will be used.

The sample size calculation revealed that 62 participants were required to ensure that a 30% decrease in the incidence of postoperative maternal hypothermia will be detected (power = 0.9 ; α= 0,05). The investigators decided to enroll 70 women because of the risks of secondary exclusions and of lost of follow up.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women

* without any major co-morbidity (ASA status 1 or 2),
* with normal singleton pregnancy,
* who will deliver by scheduled caesarean section under spinal anesthesia at gestational age ≥ 37 weeks of amenorrhea,
* Aged ≥ 18 years
* with health insurance

Exclusion Criteria:

* Patient refusal to participate in the study
* Maternal temperature ≥38.0 ° C or <36.0 ° C at the time of randomization,
* Spinal anaesthesia refused or contraindicated,
* unplanned caesarean section
* caesarean delivery scheduled since less than 48 hours
* caesarean section performed under epidural or general anesthesia
* participation of the mother in another interventional research or intervention, or during the exclusion period following a previous search
* unability to give written consent
* body mass index> 40kg / m2
* gravidic hypertensive disease
* uncontrolled diabetes
* cardiovascular disease under treatment
* coagulation disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Maternal postoperative hypothermia | until Hour 12
  Obtained by placing a skin sensor on the right temporal region and measured using the 3M™ SpotOn™ Monitoring System on arrival at the PACU Hypothermia is defined as a Temperature <36°C

SECONDARY OUTCOMES:
Maternal Shivering | Until Hour 12
  Measured on a 4 points scale (0 = no chills, 1 = intermittent, low intensity, 2 = moderate, 3 = continuous) Just before the spinal anesthesia and every 10 minutes in the operative room
Maternal shivering | Until Hour 12
  Score of 4 points (0 = no chills, 1 = intermittent, low intensity, 2 = moderate, 3 = continuous and intense) On arrival at SSPI, one hour and 2 hours after, and just before leaving the PACU
Maternal Thermal discomfort | until Hour 12
  Visual analogic scale between 0 and 100 (0: absence of thermal discomfort, 100: extreme thermal discomfort) Just before the spinal anesthesia and every 10 min during the surgery
Maternal Thermal discomfort | Until Hour 12
  Numerical scale between 0 and 100 (0: absence of thermal discomfort, 100: extreme thermal discomfort) On arrival at SSP, one hour and 2 hours after, and just before leaving the PACU
Need of active maternal warming | Until Hour 12
  use of a air forced warming blanked, peroperatively and Until H2 after surgery
Neonatal core hypothermia | Within 30th minutes of life
  Measure of Temperature °C with cutaneous thermometer
Apgar score | minute 1 after birth
  Clinically evaluated
Apgar score | minute 5 after birth
  Clinically evaluated
Apgar score | minute 10 after birth
  Clinically evaluated :assessment of the newborn infant well-being
Arterial umbilical pH measurement (physiological parameter) | Within 30th minutes of life
  Blood test
Arterial umbilical base deficit measurement | Within 30th minutes of life
  Blood test
Variation in perioperative hemoglobinemia | Within 24hours before cesarean and one day after surgery
  Blood test
Hemoglobin concentration | one day after surgery
  blood test
Postpartum anemia | One day after surgery
  Maternal hemoglobin concentration
Maternal postoperative recovery | between day 3 and day 5 after surgery
  6-minute walk test (6 MWT)
Estimation of Quality of life | at the time of the postoperative appointment, around 40 days after surgery
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Pierre Bonnet, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Pascal Alfonsi, Principal Investigator — Saint Joseph Hospital, Paris
Locations (1):
- Cochin Hospital, Port-Royal Maternity, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sessler DI. Complications and treatment of mild hypothermia. Anesthesiology. 2001 Aug;95(2):531-43. doi: 10.1097/00000542-200108000-00040. No abstract available. PMID 11506130
- [Background] Perlman J, Kjaer K. Neonatal and Maternal Temperature Regulation During and After Delivery. Anesth Analg. 2016 Jul;123(1):168-72. doi: 10.1213/ANE.0000000000001256. PMID 27314693
- [Background] Butwick AJ, Lipman SS, Carvalho B. Intraoperative forced air-warming during cesarean delivery under spinal anesthesia does not prevent maternal hypothermia. Anesth Analg. 2007 Nov;105(5):1413-9, table of contents. doi: 10.1213/01.ane.0000286167.96410.27. PMID 17959975
- [Background] Horn EP, Bein B, Steinfath M, Ramaker K, Buchloh B, Hocker J. The incidence and prevention of hypothermia in newborn bonding after cesarean delivery: a randomized controlled trial. Anesth Analg. 2014 May;118(5):997-1002. doi: 10.1213/ANE.0000000000000160. PMID 24681658
- [Background] Yokoyama K, Suzuki M, Shimada Y, Matsushima T, Bito H, Sakamoto A. Effect of administration of pre-warmed intravenous fluids on the frequency of hypothermia following spinal anesthesia for Cesarean delivery. J Clin Anesth. 2009 Jun;21(4):242-8. doi: 10.1016/j.jclinane.2008.12.010. Epub 2009 Jun 6. PMID 19502035
- [Background] Sultan P, Habib AS, Cho Y, Carvalho B. The Effect of patient warming during Caesarean delivery on maternal and neonatal outcomes: a meta-analysis. Br J Anaesth. 2015 Oct;115(4):500-10. doi: 10.1093/bja/aev325. PMID 26385660
- [Background] Cobb B, Cho Y, Hilton G, Ting V, Carvalho B. Active Warming Utilizing Combined IV Fluid and Forced-Air Warming Decreases Hypothermia and Improves Maternal Comfort During Cesarean Delivery: A Randomized Control Trial. Anesth Analg. 2016 May;122(5):1490-7. doi: 10.1213/ANE.0000000000001181. PMID 26895002